CLINICAL TRIAL: NCT02501304
Title: Feasibility Study of the ReVENT Sleep Apnea System for the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: Feasibility Study of the ReVENT Sleep Apnea System
Acronym: REV-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revent Medical International B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REV-001
Record Dates: First submitted 2015-07-14; First posted 2015-07-17 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReVENT Sleep Apnea System (Experimental): All patients will be implanted with the ReVENT Sleep Apnea System
  Interventions: Device: ReVENT Sleep Apnea System

INTERVENTIONS:
Device: ReVENT Sleep Apnea System — The ReVENT Sleep Apnea System consists of minimally invasive biocompatible devices that are placed into the tongue base and palate of patients with obstructive sleep apnea

SUMMARY:
This is a prospective, multi-center, single arm, feasibility study to evaluate the safety and effectiveness of the ReVENT Sleep Apnea System for the treatment of Obstructive Sleep Apnea.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OSA with AHI 15-40
* Body Mass Index (BMI) ≤ 32
* Refused or failed Continuous Positive Airway Pressure (CPAP)
* Evidence of airway collapse at soft palate and/or base of tongue

Exclusion Criteria:

* Prior OSA surgery
* Anatomy unable to accommodate implants
* Chronic immunosuppressive therapy or known problems with wound healing
* Type I or II diabetes
* Active systemic infection
* Pregnancy
* Other major medical conditions that could confound outcome measures or interfere with study completion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2013-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 24 months post-procedure
  Decrease in polysomnographically measured AHI post-intervention compared to baseline

IPD SHARING:
Plan to Share IPD: Yes